CLINICAL TRIAL: NCT03009201
Title: A Phase 1B Study of Ribociclib in Combination With Doxorubicin in Advanced Soft Tissue Sarcomas
Brief Title: Ribociclib and Doxorubicin in Treating Patients With Metastatic or Advanced Soft Tissue Sarcomas That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lara Davis, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016070; NCI-2016-01794 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016070 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2016-12-05; First posted 2017-01-04 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Advanced Soft Tissue Sarcoma; Locally Advanced Angiosarcoma; Locally Advanced Leiomyosarcoma; Locally Advanced Liposarcoma; Locally Advanced Malignant Peripheral Nerve Sheath Tumor; Locally Advanced Myxofibrosarcoma; Locally Advanced Undifferentiated Pleomorphic Sarcoma; Metastatic Angiosarcoma; Metastatic Epithelioid Sarcoma; Metastatic Fibrosarcoma; Metastatic Liposarcoma; Metastatic Malignant Peripheral Nerve Sheath Tumor; Metastatic Myxofibrosarcoma; Metastatic Soft Tissue Sarcoma; Metastatic Synovial Sarcoma; Metastatic Undifferentiated Pleomorphic Sarcoma; Myxofibrosarcoma; Pleomorphic Rhabdomyosarcoma; Stage III Soft Tissue Sarcoma AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7; Undifferentiated (Embryonal) Sarcoma; Unresectable Leiomyosarcoma; Unresectable Liposarcoma; Unresectable Malignant Peripheral Nerve Sheath Tumor; Unresectable Soft Tissue Sarcoma; Unresectable Synovial Sarcoma; Unresectable Undifferentiated Pleomorphic Sarcoma
MeSH Terms: conditions — Hemangiosarcoma; Sarcoma; Fibrosarcoma; Liposarcoma; Neurofibrosarcoma; Dermatofibrosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Disorders of Sex Development | interventions — Doxorubicin; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ribociclib, doxorubicin hydrochloride) (Experimental): Patients receive ribociclib PO daily on days 1-7, and doxorubicin hydrochloride IV on day 10. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive ribociclib PO daily on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Ribociclib

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011

SUMMARY:
This phase Ib trial studies the side effects and best dose of ribociclib when giving together with doxorubicin hydrochloride in treating patients with soft tissue sarcomas that has spread to other places or that cannot be removed by surgery (advanced). Ribociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ribociclib and doxorubicin hydrochloride may work better in treating patients with soft tissue sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase 2 dose (RP2D) of ribociclib in combination with doxorubicin in subjects with advanced soft tissue sarcomas.

SECONDARY OBJECTIVES:

I. To assess preliminary anti-tumor activity of ribociclib in combination with doxorubicin in subjects with advanced soft tissue sarcomas.

II. To characterize the safety and tolerability of ribociclib in combination with doxorubicin.

OUTLINE: This is a dose-escalation study of ribociclib.

Patients receive ribociclib orally (PO) daily on days 1-7, and doxorubicin hydrochloride intravenously (IV) on day 10. Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients without disease progression after 6 cycles receive ribociclib PO daily on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up within 30 days and then every 12 weeks for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of intermediate or high-grade soft tissue sarcoma for which single-agent doxorubicin is appropriate therapy, including but not limited to:

  * Synovial sarcoma
  * Fibrosarcoma
  * Undifferentiated sarcoma
  * Liposarcoma
  * Leiomyosarcoma
  * Angiosarcoma
  * Malignant peripheral nerve sheath tumor
  * Pleomorphic rhabdomyosarcoma
  * Myxofibrosarcoma
  * Epithelioid sarcoma
  * Undifferentiated pleomorphic sarcoma
* Locally advanced unresectable or metastatic disease with no standard curative therapy available
* Archival tumor tissue retinoblastoma-associated protein (pRb) positive by immunohistochemistry (IHC)
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* All races and ethnic groups will be included; for subjects between the ages of 12-18 years only, body surface area (BSA) must be >= 1.28 m^2
* Ejection fraction of >= 50% by echocardiogram or multi-gated acquisition (MUGA) scan
* Female subjects of childbearing potential must have a negative urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at time of screening and within 14 days prior to planned first dose of ribociclib
* Willing to use adequate contraception throughout the study and for 3 weeks after study drug discontinuation
* Meets the following standard 12-lead electrocardiography (ECG) parameters at screening (defined as the mean of the triplicate ECGs; ECGs done in triplicate do not have a defined interval between assessments):

  * Corrected QT using Fridericia's correction formula (QTcF) interval at screening < 450 msec for males and < 470 msec for females (using Fridericia's correction)
  * Resting heart rate =< 100 beats per minute (bpm)
* Absolute neutrophil count (ANC) >= 1.5 K/cu mm
* Platelets (no transfusion within prior 7 days) >= 100 K/cu mm
* Hemoglobin (no transfusion within prior 7 days) >= 9.0 g/dL
* Total bilirubin < institutional upper limit of normal (ULN), except for subjects with documented Gilbert's syndrome, for which =< 3.0 x ULN or direct bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT) in the absence of liver metastases: =< 2.5 x ULN; if the subject has liver metastases: < 5 x ULN
* Serum creatinine < 1.7 mg/dL
* Potassium within institutional normal limit (WNL)
* Corrected calcium WNL
* Magnesium WNL
* International normalized ratio (INR) =< 1.5

  * Use of rivaroxaban, apixaban, edoxaban or warfarin is an exclusion criteria; therapy with heparin, low molecular weight heparin (LMWH), dabigatran or fondaparinux is allowed
* All prior treatment-related toxicities resolved to =< grade 1 or are determined to be clinically stable by the investigator
* Has completed prior therapies according to the criteria below:

  * Cytotoxic chemotherapy - at least 21 days since last dose prior to first dose of ribociclib
  * Small molecule inhibitors - at least 14 days since last dose prior to first dose of ribociclib
  * Monoclonal antibodies - at least 3 half-lives since last dose prior to first dose of ribociclib; exception: denosumab for bony metastases is allowable
  * Immunotherapy (e.g. tumor vaccines) - at least 42 days since last dose prior to first dose of ribociclib
  * Radiation - at least 14 days since last dose prior to first dose of ribociclib
* Able to swallow capsules
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy > 3 months
* Ability to understand and the willingness to sign a written informed consent document; subject has signed the informed consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirements

Exclusion Criteria:

* Subjects with low grade tumors (histologic grade 1/3)
* Histologic diagnosis for which single-agent doxorubicin is NOT appropriate therapy, including but not limited to:

  * Alveolar or embryonal rhabdomyosarcoma
  * Ewings sarcoma or primitive neuroectodermal tumor (PNET)
  * Osteosarcoma
  * Gastrointestinal stromal tumor (GIST)
* Prior systemic therapy with an anthracycline for any indication
* Known hypersensitivity to any of the excipients of ribociclib or doxorubicin (including to peanut and soy)
* Currently receiving any of the following that cannot be discontinued at least 7 days prior to starting study drug:

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
  * Medications with a narrow therapeutic window that are predominantly metabolized through CYP3A4/5
  * Herbal supplements, such as St. John's wort; the use of marijuana or its derivatives is allowed in States with statutes permitting the use of recreational or medical marijuana
* Uncontrolled intercurrent medical condition including, but not limited to:

  * Uncontrolled infection
  * Symptomatic congestive heart failure (New York Heart Association [NYHA] class III-IV)
  * Acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  * Uncontrolled cardiac arrhythmia or arrhythmia requiring medication other than beta blocker
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, etc.)
* Concurrent malignancy or malignancy within 3 years prior to starting study drug, except:

  * Malignancies that have completed therapy and are considered by their physician to be at less than 30% risk of relapse, or
  * Malignancies not requiring treatment (e.g., RAI stage 0 chronic lymphocytic leukemia [CLL])
* Central nervous system (CNS) involvement unless they meet ALL of the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
  * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea/vomiting/diarrhea, malabsorption syndrome, or major small bowel resection)
* Known history of human immunodeficiency virus (HIV) infection (testing not mandatory); NOTE: HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with ribociclib; in addition, these subjects are at increased risk of lethal infections when treated with marrow suppressive therapy; appropriate studies will be undertaken in subjects receiving combination antiretroviral therapy when indicated
* Systolic blood pressure (SBP) > 160 mmHg or < 90 mmHg at screening; if initial screening SBP is outside of the eligible range, blood pressure may be re-checked after intervention; SBP must be documented as stable and within the eligible range prior to starting study drug
* Currently receiving rivaroxaban, apixaban, endoxaban, warfarin or other warfarin derived anticoagulant; therapy with heparin, low molecular weight heparin (LMWH), dabigatran or fondaparinux is allowed; if transitioning from a prohibited anticoagulant, a minimum washout of 7 days from last dose of the prohibited medication is required prior to ribociclib start
* Participation in a prior investigational interventional study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
* Major surgery within 14 days prior to starting study drug or has not recovered from surgical complications (tumor biopsy is not considered as major surgery)
* History of congenital long QT syndrome or torsades de pointes
* History of non-compliance to medical regimen or inability to grant consent
* Pregnant or nursing (lactating) women; breastfeeding should be discontinued

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) of adverse events | Up to 21 days
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.03. All adverse events (AEs) will be tabulated and summarized by major organ category, grade, anticipation, and drug attribution. Serious adverse events (SAE) specific incidence and exact 95% confidence interval will be provided where appropriate.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From first dose of protocol therapy to time of documented radiographic and/or clinical disease progression or death from any cause, whichever occurs first, assessed up to 12 months
  The Kaplan-Meier product limit method will be used to estimate PFS of the median PFS and PFS rates at clinically relevant time points will be provided with the 90% confidence interval (CI).
Objective response rate (ORR) | Up to 12 months
  Will be defined as the proportion of patients who achieved a complete response or a partial response. Will be assessed based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1. The ORR, along with exact two-sided 95% confidence intervals, will be reported for the study.
Incidence of adverse events, SAEs | Up to 12 months
  Will be assessed by NCI CTCAE v 4.03. Analyses will be performed for all patients having received at least one dose of study drug. Serious adverse events, AEs will be summarized using descriptive statistics.
Incidence of dose modifications (interruptions, reductions, intensity) due to adverse events | Up to 12 months
  Analyses will be performed for all patients having received at least one dose of study drug. AEs leading to withdrawal/dose interruptions/dose modification will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Lara E Davis, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States